CLINICAL TRIAL: NCT03392103
Title: Adjuvant IMRT With Concommitant Raltitrexed Chemotherapy for Locally Advanced Gastric Cancer After D0/D1 Radical Resection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, Zhou Fuxiang, Principal Investigator, Clinical Professor, Zhongnan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCCSC G03
Record Dates: First submitted 2017-12-19; First posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: Gastric Cancer
Keywords: Raltitrexed; IMRT
MeSH Terms: conditions — Stomach Neoplasms | interventions — raltitrexed; Radiotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- postoperative CRT (Experimental): postoperative CRT: Treatment including postoperative radiotherapy (IMRT) with concurrent chemotherapy of Raltitrexed. Radiotherapy will be delivered to a planning target volume with a dose of 45-50.4Gy (1.8-2.0Gy daily) using with Intensity-Modulated Radiotherapy technique. During the radiation treatment, concurrent chemotherapy will be delivered (Raltitrexed, intravenous infusion, 3 mg/m2, on w1 and w4).
  Interventions: Drug: Raltitrexed; Radiation: postoperative radiotherapy

INTERVENTIONS:
Drug: Raltitrexed — concurrent chemotherapy
  Other Names: Raltitrexed Injectable Solution
Radiation: postoperative radiotherapy — concurrent postoperative radiation therapy
  Other Names: adjuvant radiotherapy

SUMMARY:
The purpose of this study is to determine whether raltitrexed concurrent with IMRT is safe, tolerable and effective in the treatment for patients with local-advanced gastric cancer after D0/D1 radical resection.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent signed.;
2. Age: 18-70 years old, sex is not restricted;
3. Pathologically diagnosed as gastric adenocarcinoma or gastroesophageal junction adenocarcinoma; did not receive neoadjuvant chemotherapy or radiotherapy before surgery;received the 2-3 cycles of chemotherapy of FOLFOX regimens or 1-2 cycles of XeLOX or SOX regimens after operation;
4. Received D0 or D1 operation, no tumor residual (R0);
5. Postoperative pathological stage of pT3N0, pT4N0 or any T, N1-2, without distant metastatic disease;
6. ECOG 0-2;
7. Normal blood analysis: WBC≥3.5 X 109/L, GRAN≥2.0 X 109/L = 2, Hb≥90g/L, PLT≥100 X 109/L;
8. Liver function: ALT or AST is less than or equal to 2.5 times of the normal high value (ULN); bilirubin is less than 1.5*ULN, serum APK is less than 2.5 * ULN;
9. Renal function: serum creatinine is less than 1.5 * ULN, and creatinine clearance rate is more than 60ml/min;
10. No previous chemotherapy or radiation therapy history;
11. No organ transplant history;
12. Urine pregnancy test results are negative for women of childbearing age in the first 7 days and not in lactation before treatment;
13. Men and women of childbearing age agreed to adopt reliable methods of contraception for 30 days before , during and after the course of the study

Exclusion Criteria:

1. Received D2 radical operation;
2. Tumor residual (R1/R2);
3. There was found evidence of distant metastasis (M1) or suspicious metastasis after examination;
4. Other cancer history, except skin basal cell carcinoma or cervix in-situ carcinoma;
5. Previously received chemotherapy or other systemic anticancer therapy, including cytotoxic drugs, targeted drugs; or had received abdominal radiotherapy;
6. Anticipate other clinical trials in four weeks before enrollment.
7. Severe complication, such as acute myocardial infarction in 6 months, uncontrolled diabetes, severe cardiac arrhythmia, etc.
8. Drug abuse history or alcohol addiction;
9. Active infection existed.
10. with severe malnutrition or severe anemia;
11. Human immunodeficiency virus (HIV) infection;
12. Pregnancy (confirmed by serum or urine beta -HCG test) or during lactation;
13. Can not tolerate this study or may be allergic to the drug used in this study;
14. Persons who have no or restricted capacity for civil conduct; or have mental illness, whom the researchers believe can not fully understand the possible complications of this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The ratio of patients occured Grade 3 or higher adverse events | From the first day of the concurrent chemoradiotherapy (CRT) to the 180th day after CRT.

SECONDARY OUTCOMES:
2-year local-regionally recurrence rate | 2 year
  The probability of locally and/or regionally recurrence at 2 year after CRT on imaging or pathological examination.
3-year local-regionally recurrence rate | 3 year
  The probability of locally and/or regionally recurrence at 3 year after CRT on imaging or pathological examination.
2-year disease-free survival probability | 2 year
  The probability of staying free from recurrence at 2 year after CRT on imaging or pathological examination.
3-year disease-free survival probability | 3 year
  The probability of staying free from recurrence at 3 year after CRT on imaging or pathological examination.
2-year overall survival probability | 2 year
  The probability of staying alive at 2 year after CRT.
3-year overall survival probability | 3 year
  The probability of staying alive at 3 year after CRT.

CONTACTS AND LOCATIONS:
Overall Officials: Fuxiang Zhou, M.D., Study Chair — Zhongnan Hospital
Locations (1):
- Zhongnan Hopital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No